CLINICAL TRIAL: NCT03022968
Title: Tau Brain Imaging in Typical and Atypical Alzheimer's Disease (AD)
Acronym: TEPTAU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PHAO14-CH/TEPTAU
Record Dates: First submitted 2017-01-09; First posted 2017-01-18 (Estimated); Last update posted 2022-09-09 (Actual); Status verified 2019-05

CONDITIONS: Alzheimer Disease; Benson's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alzheimer disease (Experimental): [18F]T807 PET
  Interventions: Drug: [18F]T807 PET
- Benson disease (Experimental): [18F]T807 PET
  Interventions: Drug: [18F]T807 PET
- Healthy volunteer (Experimental): [18F]T807 PET
  Interventions: Drug: [18F]T807 PET

INTERVENTIONS:
Drug: [18F]T807 PET — Imaging with [18F]T807 PET

SUMMARY:
Recently revised Alzheimer Disease (AD) diagnostic1described nonamnestic presentations: 1/ language presentation (logopenic progressive aphasia) 2/ visuospatial presentation (posterior cortical atrophy or PCA) and 3/ executive dysfunction. AD pathological changes may precede the clinical diagnosis of dementia of AD type for a while2. Biomarkers have been developed: biomarkers of brain amyloid-beta (Aß) (CerebroSpinal Fluid CSF concentration ßamyloid, molecular imaging with amyloid targeted PET ligands), biomarkers of neural degeneration (MRI hippocampal volume, regional metabolism as assessed by PET with [18F]-FDG) and may be used to made early detection of the neuropathology associated with AD Even if CSF biomarkers (tau, p-tau and β amyloïd are interesting to improve diagnosis of AD, they cannot provide topographic information. PET tau imaging seems to be promise to evaluate quantitative and spatial assessment of tau lesions both in AD and fronto-temporal lobar dementia.

The hypothesis of the research is that it exists a different regional pattern of tracer retention across brain regions according to clinical symptoms : temporal for logopenic aphasia and occipital for posterior cortical atrophy.

ELIGIBILITY:
Inclusion Criteria:

* 50 years old and more
* native langage: french
* study level upper (or equal) than 7 year (considering first year of grammar-school as start)
* correct sensory abilities (auditive device allowed) for tests
* affiliation to social security
* Informed, written consent form
* for Alzheimer disease group: people with Alzheimer Disease defined as National Institute of Neurological and Communicative Disorders and Stroke (NINCDS) and the Alzheimer's Disease and Related Disorders Association (ADRDA) standards: Light to mild AD defined by Mini-Mental State Examination (MMSE) score between 15 and 25 (included)
* for Benson disease group: Benson disease following Mendez et al (2002) and Tang Wai et al (2004) criteria
* for healthy volunteer group: normal MMS score (more than 26 for bachelor level)

Exclusion Criteria:

* history of disease with consequances on cognitive functioning (tumor, stroke, head trauma, etc.), cerebral surgery
* use of alchohol and/or drug
* anormalies in neurological exam (focal deficit) not included in the classic symptoms
* contraindication to magnetic resonance imaging (RMI)
* contraindication to PET: people with prolongation of QT interval or taking medication that can lead to "torsades de pointe".
* claustrophobia
* person with legal protection
* exclusion period because of participation to another experimental protocol and actual participation to an experimental protocol
* pregnant or lactating woman or able to procreate and without contraception

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Tau density on PET imaging | 3 months
  density pattern of aggregated tau using tau targeting PET imaging with [18F]-T807, in Standardized uptake value (SUV)
Tau distribution on PET imaging | 3 months
  distribution pattern of aggregated tau using tau targeting PET imaging with [18F]-T807, in Standardized uptake value (SUV)

SECONDARY OUTCOMES:
p-tau CSF biomarkers | inclusion
  p-tau dosing in pg/mL
βamyloid CSF biomarkers | inclusion
  βamyloid dosing in pg/mL
Cognitive profile with Hamilton depression scale (MADRS) | inclusion
  neuropsychological score of Hamilton depression scale (MADRS) on 30 points.
Cognitive profile with Mini mental state evaluation (MMSE) | inclusion
  neuropsychological score of Mini mental state evaluation (MMSE) on 60 points

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No